CLINICAL TRIAL: NCT01181466
Title: A Study of the AeriSeal® System Administered at 3 to 4 Sites During a Single Treatment Session for Lung Volume Reduction in Patients With Advanced Emphysema
Brief Title: AeriSeal® System for Lung Volume Reduction in Patients With Advanced Emphysema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-C10-002PLV
Record Dates: First submitted 2010-07-13; First posted 2010-08-13 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Emphysema; COPD; Lung Diseases
Keywords: PLVR; BLVR; AeriSeal; treatment; device; breathing; COPD; emphysema; polymeric lung volume reduction; biologic lung volume reduction; heterogeneous; homogeneous; Pathologic Processes; Respiratory Tract Diseases; Lung Diseases; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Aspiration; Emphysema; Pathologic Processes; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AeriSeal System — The AeriSeal System will be Administered at 3 to 4 Pulmonary Subsegments During a Single Treatment session.

SUMMARY:
The purpose of this study is to assess the procedural and post-procedural safety and efficacy of AeriSeal therapy at up to 4 subsegments during a single treatment session in patients with GOLD Stage III/IV homogeneous or heterogeneous emphysema.

DETAILED DESCRIPTION:
Emphysema is a progressive, debilitating disease characterized by destruction of lung tissue as a result of inflammation caused by exposure to noxious inhaled agents for extended periods. The most common cause of this condition is cigarette smoking, although genetic, occupational, and environmental causes account for up to 10% of cases. Despite aggressive public health initiatives aimed at discouraging the use of cigarettes, smoking-related lung diseases remain a significant cause of disability and death worldwide. Due to the number of current and new smokers, emphysema is expected to remain a leading cause of morbidity and mortality for years to come.

The AeriSeal System is a novel device system being developed for the treatment of advanced emphysema. The AeriSeal System is administered bronchoscopically, and designed to provide the physiological benefits of lung volume reduction without the risks and cost of major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of advanced emphysema as defined by FEV1/FVC<70% predicted, FEV1 of <50% predicted, TLC > 100% predicted, and RV > 135% predicted.
* Patients must have persistent symptoms despite medical therapy and either not be candidates for Lung Volume Reduction Surgery (LVRS) or have elected not to undergo LVRS.
* Patients must be > 40 years of age, have symptoms despite medical therapy, and have none of the prespecified co-morbid conditions that could influence study outcomes or their ability to tolerate bronchoscopy.

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in Percent Volume of Lung | 12 weeks following treatment
  Computed Tomography (CT) evidence of lobar volume reduction at site(s) of AeriSeal Foam Sealant administration at 12 weeks post treatment, assessed quantitatively by digital integration of CT dicom images collected using a standardized image acquisition and reconstruction algorithm.

SECONDARY OUTCOMES:
Change in the ratio of Residual Volume (RV) to Total Lung Capacity (TLC) | 12 weeks following treatment
  Change from baseline at 12 weeks in RV/TLC
Change in Forced Expiratory Volume in 1 Second (FEV1) | 12 weeks following treatment
  Change from baseline at 12 weeks in FEV1
Change in Forced Vital Capacity (FVC) | 12 weeks following treatment
  Change from baseline at 12 weeks in FVC
Change in distance walked in six minutes | 12 weeks following treatment
  Change from baseline at 12 weeks in 6 Minute Walk Test (6MWT)
Change in Medical Research Council Dyspnea (MRCD) score | 12 weeks following treatment
  Change from baseline at 12 weeks in MRCD score
Change in St. George's Respiratory Questionnaire (SGRQ) domain score | 12 weeks following treatment
  Change from baseline at 12 weeks in SGRQ total domain score

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - The Soroka Medical Center, Beersheba
  - The Rabin Medical Center, Petah Tikva

REFERENCES:
- [Derived] Magnussen H, Kramer MR, Kirsten AM, Marquette C, Valipour A, Stanzel F, Bonnet R, Behr J, Fruchter O, Refaely Y, Eberhardt R, Herth FJ. Effect of fissure integrity on lung volume reduction using a polymer sealant in advanced emphysema. Thorax. 2012 Apr;67(4):302-8. doi: 10.1136/thoraxjnl-2011-201038. Epub 2012 Feb 28. PMID 22374920
- See also: Aeris Therapeutics — http://www.aerist.com/